CLINICAL TRIAL: NCT03767114
Title: Estimation of Level of ERAP1 Expression in Lesional and Non Lesional Skin of Psoraitic Patients and Healthy Controls.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Rana F Hilal, MD, Lecturer of dermatology, Kasr El Aini Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: EgyERAP
Record Dates: First submitted 2018-12-05; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-12

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cases of psoriasis (Experimental): group of 25 cases of psoriasis subjected to skin biopsy for detection of lesional and non lesional expression of ERAP1 by RT-PCR
  Interventions: Diagnostic Test: RT-PCR for ERAP1 detection
- normal controls (Experimental): group of 30 age and sex matched healthy controls o subjected to skin biopsy from normal skin for detection of expression of ERAP1 by RT-PCR
  Interventions: Diagnostic Test: RT-PCR for ERAP1 detection

INTERVENTIONS:
Diagnostic Test: RT-PCR for ERAP1 detection — Reverse transcriptase -Polymerase Chain Reaction for ERAP1 detection

SUMMARY:
A 4mm Punch biopsy is obtained from lesional and non lesional skin of 25 psoraitic patients as well as of 30 controls.

Skin biopsy from patients (psoriasis lesional and non lesional) & control will be kept in lysis solution (which contains RNAase inhibitor) for the stability of the parameter to be assessed. ERAP-1 gene expression will Research Template 5 Final Version: 8/3/2 016 be detected by quantitative real time -PCR, which include RNA extraction, cDNA synthesis & PCR.

ELIGIBILITY:
Inclusion Criteria:

* patients with psoriasis vulgaris
* patients over 18 years of age
* both sexes

Exclusion Criteria:

* patients on treatment for psoriasis within the last two months
* assoiciated autoimmune diseases eg SLE
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Estimation of lesional ERAP1 in psoriatic skin | Maximum 2 years
  DPCRetection of level of expression of ERAP 1 in lesional skin of psoriasis patients by RT-

SECONDARY OUTCOMES:
Estimation of non lesional ERAP1 in psoriatic skin | Maximum 2 years
  Detection of level of expression of ERAP 1 in non lesional skin of psoriasis patients by RT-PCR.